CLINICAL TRIAL: NCT02361983
Title: Airway Management in Thoracic Surgery and Incidence Rate of Dislocation and Related Intraoperative Hypoxemia: State of the Art in Italy
Brief Title: Airway Management in Thoracic Anesthesia in Italy
Acronym: AIRTHOR
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Giorgio Della Rocca, Professor and Chair of Anesthesia and Intensive Care Medicine Medical School of the University of Udine University of Udine. Udine, Italy, Azienda Ospedaliera S. Maria della Misericordia
Other Study IDs: AirwaysThor; Local ethics committee ALI01 (Other: AOU Santa Maria della Misericordia)
Record Dates: First submitted 2012-12-03; First posted 2015-02-12 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DLT: Patients managed with a Double lumen tube (DLT)
  Interventions: Device: Double lumen tube
- Bronchial blockers: Patients managed with a Bronchial blocker (BB)
  Interventions: Device: Bronchial blocker

INTERVENTIONS:
Device: Double lumen tube — Patients managed with a double lumen tube for one lung ventilation
  Other Names: DLT
  Groups: DLT
Device: Bronchial blocker — Patients managed with a bronchial blocker for one lung ventilation
  Other Names: BB
  Groups: Bronchial blockers

SUMMARY:
The aim of this study is to evaluate the positioning time and the malpositioning rate of DLTs and BBs, the degree of difficulty perceived in device positioning, the use of bronchoscopy (BRO), and the quality of lung collapse achieved during ONE LUNG VENTILATION.

DETAILED DESCRIPTION:
Safety and efficacy of the double-lumen tubes (DLT) and bronchial blockers (BB) for lung isolation in patients undergoing thoracic surgery have been extensively studied and most of the results show similar rates of successful placement and lung collapse. DLT and BB are more frequently inserted by anesthetists who are expert in thoracic anesthesia, with dedicated but different training.

The first objective of this study was to evaluate the positioning time and the malpositioning rate of DLTs and BBs, the degree of difficulty perceived in device positioning, the use of bronchoscopy (BRO), and the quality of lung collapse achieved during OLV.

A prospective observational study was designed. To check the optimal DLT (Broncho-Cath Covidien, Ireland, Dublin, Teleflex Medical, Athlone, Irelanad) and/or BB (Uniblocker, Phycon, Fuji, Japan Arndt Cohen Cook, Australia), placement a fiberoptic bronchoscope (FOB) was used. The lung collapse was assessed by surgeons.

Time from laringoscopy to the correct placement of the device, confirmed with FOB, was checked.

Data were analyzed with Student't Test and Chi-square test; p value < 0.05 was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* patients who need one lung ventilation undergoing thoracic surgery

Exclusion Criteria:

* age < 18 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 2225 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
DOUBLE LUMEN TUBE AND BRONCHIAL BLOCKER POSITIONING SUCCESS RATE: RESIDENTS vs. ATTENDING ANESTHETISTS. | 11/19/2012
  A prospective randomized trial was designed. To check the optimal DLT (Broncho-Cath Covidien, Ireland, Dublin, Teleflex Medical, Athlone, Irelanad) and/or BB (Uniblocker, Phycon, Fuji, Japan Arndt Cohen Cook, Australia), placement a fiberoptic bronchoscope (FOB) was used. The lung collapse was assessed by surgeons.
  Time from laringoscopy to the correct placement of the device, confirmed with FOB, was checked.
  Data were analyzed with Student't Test and Chi-square test; p value < 0.05 was considered to be significant.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Della Rocca, prof, Principal Investigator — AOU Santa maria della Misericordia
Locations (1):
- Department of Anesthesia and Intensive Care, Udine, Udine/Italy, Italy

REFERENCES:
- [Background] Narayanaswamy M, McRae K, Slinger P, Dugas G, Kanellakos GW, Roscoe A, Lacroix M. Choosing a lung isolation device for thoracic surgery: a randomized trial of three bronchial blockers versus double-lumen tubes. Anesth Analg. 2009 Apr;108(4):1097-101. doi: 10.1213/ane.0b013e3181999339. PMID 19299767
- [Background] Campos JH, Hallam EA, Ueda K. Training in placement of the left-sided double-lumen tube among non-thoracic anaesthesiologists: intubation model simulator versus computer-based digital video disc, a randomised controlled trial. Eur J Anaesthesiol. 2011 Mar;28(3):169-74. doi: 10.1097/EJA.0b013e328340c332. PMID 21088594